CLINICAL TRIAL: NCT01833351
Title: Pharmacokinetic Evaluation of Intravenous Ascorbic Acid
Brief Title: Evaluation of Intravenous Ascorbic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Jeanne Drisko, MD, CNS, FACN, Riordan Endowed Professor of Orthomolecular Medicine, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12680
Record Dates: First submitted 2012-05-30; First posted 2013-04-16 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Safety and Pharmacokinetics of Intravenous Ascorbate
Keywords: Phase I; safety and pharmacokinetics,; intravenous ascorbate,; IV Vitamin C,; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I, IV Vitamin C Healthy Normals (Experimental): Safety and pharmacokinetics of intravenous ascorbate,IV Vitamin C.
  Interventions: Drug: IV Vitamin C
- Phase 1 IV Vitamin C- Cancer Patients (Experimental): Safety and pharmacokinetics of intravenous ascorbate,IV Vitamin C.
  Interventions: Drug: IV Vitamin C

INTERVENTIONS:
Drug: IV Vitamin C — We will begin by enrolling 3 people at each dose level and if there are any problems seen, we will enroll 3 more people to that dose to see if that problem happens again and this may total a maximum of 6 people. Therefore a maximum of 6 people may be enrolled at each of these Vitamin C dose levels, 1 gram, 5 grams, 10 grams, 25 grams, 50 grams, 75 grams, and 100 grams.
  If you are eligible for the study and decide to participate, the total time involved could be approximately 4 weeks.
  Other Names: IV Ascorbate
Drug: IV Vitamin C — There will be 4 dose levels of intravenous vitamin C selected for this part of the study. The first dose level will be 25% of the top dose level found to be safe in Part 1, followed by 50% of the top dose level, followed by 75% of the top dose level, and finally 100% of the top dose. For example, if 100 grams of vitamin C given by vein is found to be safe in Part 1, then the first dose level we will choose will be 25 grams, followed by 50 grams, then 75 grams, and finally 100 grams.
  Three to 6 people will be invited to participate in each of the dose levels and you will be asked to get a total of 4 doses at that level spread out over 4 weeks. In addition, you will have an initial visit and a follow-up visit both lasting 30 minutes. This will total 6 visits.
  Other Names: IV Ascorbate

SUMMARY:
This Phase I study will be conducted in 2 parts to examine safety and pharmacokinetics of escalating doses of intravenous ascorbic acid (AA) first in healthy volunteers followed by evaluation in oncology subjects. The study will be conducted in the Program in Integrative Medicine Infusion Clinic at the University of Kansas Medical Center in conjunction with the Program in Integrative Medicine, Kansas Cancer Research Institute, Department of Pharmacy, Department of Medical Oncology, the Division of Surgical Oncology,and with consultants from the NIH, and FDA.

DETAILED DESCRIPTION:
The purpose of this study is to examine what happens when Vitamin C enters into the body, and the speed and ways it travels through the body, and the rate at which it exits the body in the urine. It is also necessary to determine if it is safe to give Intravenous Vitamin C at high doses.

ELIGIBILITY:
PART 1 ELIGIBILITY CRITERIA

Inclusion:

* Healthy adults age 21 or older
* Laboratory: ANC ≥1,500/mm3,

  * Hemoglobin > 8g/dL,
  * platelet ≥ 100,000/mm3,
  * total bilirubin ≤ 1.5 mg/dL,
  * creatinine ≤2.0 mg/dL,
  * transaminase (AST/ALT) ≤2.5X upper limit,
  * urine uric acid < 1,000mg/d,
  * urine pH <6,
  * urine oxalate <60 mg/d.
* Participants who have no language barrier, are cooperative, and can give informed consent before entering the study after being informed of the medications and procedures to be used in this study may participate.

Exclusion:

* Glucose-6-phosphate-dehydrogenase (G6PD) deficiency
* History of bleeding disorder
* History of oxalate renal calculi; urine oxalate level > 60 mg/d at baseline
* History of iron overload or hemochromatosis
* Participants with evidence of a significant psychiatric disorder by history/examination that would prevent completion of the study will not be allowed to participate.
* Co-morbid condition that would affect survival: end stage congestive heart failure, unstable angina, myocardial infarction within 6 weeks of study, uncontrolled blood sugars ≥ 300 mg/dL, participants with known chronic active hepatitis or cirrhosis.
* Participants who consume an excess of alcohol or abuse drugs (an excess of alcohol is defined as more than four of any one of the following per day: 30mL distilled spirits, 340mL beer, or 120mL wine) will not be allowed.
* Participants who smoke tobacco products will not be allowed to participate.

PART 2 ELIGIBILITY CRITERIA

Inclusion:

* Oncology participants must have histologically or cytologically diagnosed malignancy.
* The oncology participants must be age 21 or older and screened for eligibility and have study approved by treating oncologist.
* Oncology participants must be unwilling or ineligible for further radiation or chemotherapy at the time of enrollment into study.
* Participants must be without evidence of active spinal cord compression and have predicted lifespan of 6-months or more.
* ECOG Performance Status 0-2

  * Eastern Cooperative Oncology Group Performance Status
  * Grade 0 = Fully active, able to carry on all pre-disease activities without restriction
  * Grade 1= Restricted in physical strenuous activity but ambulatory and able to carry out work of a light or sedentary nature e.g. light housework, office work
  * Grade 2 = Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours.
* Laboratory:

  * ANC ≥1,500/mm3,
  * Hemoglobin > 8g/dL,
  * platelet ≥ 100,000/mm3,
  * total bilirubin ≤ 1.5 mg/dL,
  * creatinine ≤2.0 mg/dL,
  * transaminase (AST/ALT) ≤2.5X upper limit,
  * urine uric acid < 1,000mg/d, urine pH <6,
  * urine oxalate <60 mg/d.
* Participants who have no language barrier, are cooperative, and can give informed consent before entering the study after being informed of the medications and procedures to be used in this study may participate.

Exclusion:

* Glucose-6-phosphate-dehydrogenase (G6PD) deficiency
* Currently receiving chemotherapy or radiation therapy
* History of bleeding disorder
* History of oxalate renal calculi; urine oxalate level > 60 mg/d at baseline
* History of iron overload or hemochromatosis
* Participants with evidence of a significant psychiatric disorder by history/examination that would prevent completion of the study will not be allowed to participate.
* ECOG Performance Status of 3-4

  * Grade 3 = Capable of only limited self care, confined to bed or chair more than 50% of waking hours.
  * Grade 4 = Completely disabled. Cannot carry on any self care. Totally confined to bed or chair) and in terminal stages of disease.
* Co-morbid condition that would affect survival: end stage congestive heart failure, unstable angina, myocardial infarction within 6 weeks of study, uncontrolled blood sugars ≥ 300 mg/dL, participants with known chronic active hepatitis or cirrhosis.
* Those who consume an excess of alcohol or abuse drugs (an excess of alcohol is defined as more than four of any one of the following per day: 30mL distilled spirits, 340mL beer, or 120mL wine) will not be allowed.
* Those who smoke tobacco products will not be allowed to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
identify the maximum tolerated dose (MTD) | Change from infusion to 24 hours past infusion
  This will be accomplished by obtaining the following evaluations: toxicity graded by the NCI CTC, urinalysis pre- and post-infusion, ECG, basic metabolic panel, bicarbonate (pH surrogate marker), CBC, and osmolality.

SECONDARY OUTCOMES:
measure how the body absorbs, distributes and excretes intravenous ascorbic acid | 0,.5,1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 24 hours post-dose
  The pro-drug ascorbic acid will be administered intravenously in escalating doses of 1, 5, 10, 25, 50, 75, and 100 grams and infused over 120 minutes with sampling pre, during, and post infusion up to 24 hours in 21 healthy adults and 12 oncology participants who unable or unwilling to receive further cytoreductive therapy.
measure the biochemical and physiological effects of intravenous ascorbic | 0,.5,1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 24 hours post-dose
  The pro-drug ascorbic acid will be administered intravenously in escalating doses of 1, 5, 10, 25, 50, 75, and 100 grams and infused over 120 minutes with sampling pre, during, and post infusion up to 24 hours in 21 healthy adults and 12 oncology participants who unable or unwilling to receive further cytoreductive therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Drisko, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Chen P, Reed G, Jiang J, Wang Y, Sunega J, Dong R, Ma Y, Esparham A, Ferrell R, Levine M, Drisko J, Chen Q. Pharmacokinetic Evaluation of Intravenous Vitamin C: A Classic Pharmacokinetic Study. Clin Pharmacokinet. 2022 Sep;61(9):1237-1249. doi: 10.1007/s40262-022-01142-1. Epub 2022 Jun 25. PMID 35750958